CLINICAL TRIAL: NCT04361786
Title: Acral Cutaneous Thrombotic Vasculopathy and Covid-19 Infection: Search for Acquired Thrombophilia and Interferon-alpha Signature
Brief Title: Acral Cutaneous Thrombotic Vasculopathy and Covid-19 Infection
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Lyon Civil Hospitals - Lyon Sud Hospital Center (Unknown); University Hospital, Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0211
Record Dates: First submitted 2020-04-17; First posted 2020-04-24 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: COVID 19
Keywords: Suspected or proved Covid-19 virus infection, current or past; Chilblains; Interferon; Vasculitis
MeSH Terms: conditions — COVID-19; Chilblains; Vasculitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and skin biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Spectrum of skin lesions may arise during Covid-19 virus infection. It includes non-specific urticaria, aphtoids lesions, but also acrosyndromes, in particular suggestive of chilblains. Pathological findings showed thrombocytic lymphocytic vasculitis. Chilblains are sometimes associated with Raynaud's phenomenon or acrocyanosis. Dermatological features may present pathophysiological similarities with the inflammatory and respiratory vascular disturbances, which makes all the gravity of this disease, or even with other organs. Indeed, genetic conditions such as familial lupus chilblains, linked to a mutation of TREX1 gene, and SAVI (Sting associated vasculopathy with onset on infancy) have similar clinical presentations. In particular, SAVI associates both acral skin and lung damage, and auto-antibodies. They have recently been identified as type I interferonopathies. Hallmark is interferon signature, i.e. hyperexpression of type I interferon in the blood.

The investigators hypothesize Covid-19 may lead to similar skin involvement as in type I interferonopathies. The interferon pathway is involved in anti-viral defense. Covid-19 could cause excessive activation of this pathway. In addition, hyperactivation of the type I interferon pathway leads to modulation of the adaptive immune response. Production of autoantibodies, in particular antiphospholipid antibodies, have thrombogenic properties. Searching for acquired hemostasis disorders and high level of interferon secondary Covid-19 virus infection, could explain this new and misunderstood skin disorder. Then, targeted therapies, both treating and preventing, could be considered.

ELIGIBILITY:
Inclusion criteria:

* Chilblains or vascular abnormalities (Raynaud's phenomenon, purpura, livedo, necrosis, acrocyanosis) of the acral skin (hands, feet, nose, ears) developping during or after a proved or suspected Covid-19 infection.

Exclusion criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients seen in Covid unity in Montpellier University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Biological acquired thrombophilia | 1 day
  Searching for presence or absence of abnormal acquired thrombophilic condition as antibodies, hemostasis disturbances. Presence or absence of thrombophilic markers in the blood

SECONDARY OUTCOMES:
Overexpression of interferon type I | 1 day
  Dosing transcriptomic interferon signature in a blood sample. Presence or absence of interferon in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Didier BESSIS, PhD, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC